CLINICAL TRIAL: NCT02283801
Title: A Phase 1, Open-label Drug Interaction Study Between Eslicarbazepine Acetate 1200mg and Lamotrigine 150mg Following Multiple Doses Administrations in Healthy Male Volunteers
Brief Title: Open-label Drug Interaction Study Between Eslicarbazepine Acetate and Lamotrigine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-119
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Group A
  * Pre-treatment: 600 mg once daily dose of eslicarbazepine acetate (ESL) administered for two consecutive days;
  * Treatment 1: 1200 mg once daily dose of eslicarbazepine acetate (ESL) administered for six consecutive days
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and lamotrigine 50 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and lamotrigine 150 mg for seventeen consecutive days
  Interventions: Drug: Eslicarbazepine acetate; Drug: Lamotrigine
- Group B (Experimental): Group B
  * Pre-treatment: 50 mg once daily dose of lamotrige (LMT) administered for two consecutive days;
  * Treatment: 150 mg once daily dose of lamotrige (LMT) administered for six consecutive days;
  * Treatment 2: Concomitant doses of eslicarbazepine acetate (ESL) 1600 mg and lamotrigine 150 mg for two consecutive days
  * Treatment 3: Concomitant doses of eslicarbazepine acetate (ESL) 1200 mg and lamotrigine 150 mg for seventeen consecutive days
  Interventions: Drug: Eslicarbazepine acetate; Drug: Lamotrigine

INTERVENTIONS:
Drug: Eslicarbazepine acetate
  Other Names: ESL
Drug: Lamotrigine
  Other Names: LMT

SUMMARY:
Single centre, open-label, multiple doses, one-sequence design study in two parallel groups of healthy volunteers

DETAILED DESCRIPTION:
Single centre, open-label, multiple doses, one-sequence design study in two parallel groups of healthy volunteers: Group A: Pre-treatment with ESL, treatment with ESL and ascending doses of Lamotrigine (LMT) in last phases; Group B: Pre-treatment with LMT, treatment with LMT and ascending doses of ESL in last phases

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Male aged of at least 18 years but not older than 45 rears with a body mass índex (BMI) greater than or equal to 19 and below 30 kg/m
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance (laboratory tests are presented in section 6.1.1.3)
* Healthy according to the medical history, laboratory results and physical examination
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 1 0 cigarettes or less per day, and an ex-smoker is defined as someone who completely stopped smoking for at least 12 months before day I of thi s study The informed consent form must be signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

* Significant history of hypersensitivity to lamotrigine, eslicarbazepine, oxcarbazepine, carbamazepine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of significant heart disease or disorder according to ECG
* Presence or history of significant central nervous system disorder like convulsion or depression
* Presence or history of significant ocular disease
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cmax - the maximum plasma concentration | Group A:Day 8 and 27: within 5 minutes prior to dosing and 0.5,1,1.5,2,2.5,3,3.5,4,6,9,12,16 and 24 hours after drug administration; Group B: Day 8 and 27 within 5 minutes prior dosing and 0.25,0.5,0.75,1,1.33,1.67,2,2.5,3,4,6,9,12,16 and 24h
AUC0-t - the area under the plasma concentration-time curve from time zero to the last sampling time | Group A:Day 8 and 27: within 5 minutes prior to dosing and 0.5,1,1.5,2,2.5,3,3.5,4,6,9,12,16 and 24 hours after drug administration; Group B: Day 8 and 27 within 5 minutes prior dosing and 0.25,0.5,0.75,1,1.33,1.67,2,2.5,3,4,6,9,12,16 and 24h

SECONDARY OUTCOMES:
tmax - the time of occurrence of Cmax | Group A:Day 8 and 27: within 5 minutes prior to dosing and 0.5,1,1.5,2,2.5,3,3.5,4,6,9,12,16 and 24 hours after drug administration; Group B: Day 8 and 27 within 5 minutes prior dosing and 0.25,0.5,0.75,1,1.33,1.67,2,2.5,3,4,6,9,12,16 and 24h